CLINICAL TRIAL: NCT04735861
Title: Sintilimab Plus Bevacizumab in Patients With Recurrent/Persistent Ovarian Clear Cell Carcinoma
Brief Title: Sintilimab Plus Bevacizumab in Recurrent/Persistent Ovarian Clear Cell Carcinoma
Acronym: INOVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Union Hospital affiliated to Tongji Medical College (Unknown); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Henan Cancer Hospital (Other Government); Hubei Cancer Hospital (Other); Shengjing Hospital (Other); Anhui Provincial Cancer Hospital (Other); Zhongnan Hospital (Other); Jingzhou Central Hospital (Other); The First People's Hospital of Jingzhou (Other); Xiangyang Central Hospital (Other); Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital & Shenzhen Hospital (Unknown)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-TJ-OCCC
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Clear Cell Carcinoma
Keywords: Ovarian clear cell carcinoma; PD-1 inhibitor; Antiangiogenic therapy
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Arm (Experimental): Sintilimab 200mg iv., q3w, up to 2 years; Bevacizumab 15mg/kg iv., q3w, up to 22 cycles. Treatment is given until confirmed progression, death, unacceptable toxicity, or any other protocol-specified criterion for withdrawal, whichever occurs first.
  Interventions: Drug: Sintilimab; Drug: Bevacizumab Biosimilar IBI305

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg iv. q3w, up to 2 years.
  Other Names: IBI308
Drug: Bevacizumab Biosimilar IBI305 — Bevacizumab 15mg/kg iv. q3w, up to 22 cycles
  Other Names: IBI305

SUMMARY:
Ovarian clear cell carcinoma (OCCC) is one of the rare subtypes of ovarian cancer, yet its prognosis is extremely poor. Previous studies indicate that both bevacizumab and PD-1 inhibitor have clinical benefits for OCCC patients. And the combination of bevacizumab and PD-1 inhibitor has shown preliminary safety and clinical activity. Therefore, this study aims to investigate the potential benefit of combination therapy for patients with OCCC.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with age ≥ 18 years old and < 75 years old.
2. There must be a histological diagnosis of ovarian clear cell carcinoma. For tumors with mixed histology, at least 70% of the tumors are composed of clear cell carcinoma.
3. Patients with recurrent or persistent ovarian clear cell carcinoma must have at least one-line pretreated platinum-containing chemotherapy.
4. Patients with recurrent or persistent ovarian clear cell carcinoma must have at least one-line pretreated platinum-containing chemotherapy.
5. According to the definition of RECIST1.1, the patient must have measurable lesions. Measurable lesions are defined as:

   * There is at least one lesion that can be accurately measured in at least one dimension;
   * When measured by CT or MRI or the diameter gauge of clinical examination, each lesion must be ≥ 10 mm. When measured by chest X-ray, each lesion must be ≥ 20 mm.
   * When lymph nodes measured by CT or MRI, the short axis of the lymph nodes must be ≥ 15 mm.
6. It must be at least 4 weeks away from the last anti-tumor treatment before starting the trial treatment.
7. No administration of immune checkpoint inhibitors before.
8. Enough archived tumor tissue blocks (or at least 10 freshly cut unstained glass slides) provided for analysis.
9. ECOG performance status score ≤ 2.
10. Expected survival time > 12 weeks.
11. Adequate hematology and organ function, including:

    * hemoglobin > 9 g/dL without blood transfusion or erythropoietin in the past 14 days.
    * ANC ≥ 1.5×109/L without using granulocyte colony stimulating factor in the past 14 days.
    * PLT ≥ 9×109/L without blood transfusion in the past 14 days.
    * TBIL ≤ 1.5 ×ULN (Gilbert syndrome allows ≤ 3 × ULN).
    * ALT and AST ≤ 2.5 × ULN (if there is liver metastasis, ALT and AST ≤ 5 × ULN).
    * Serum Cr ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula).
    * Adequate coagulation function, defined as INR or PT ≤ 1.5 × ULN.
    * Normal thyroid function is defined as TSH within the normal range. If the baseline TSH is outside the normal range, patients with total T3 (or FT3) and FT4 are within the normal range can also be included.
    * Myocardial enzyme spectrum is within the normal range (patients with simple laboratory abnormalities judged by the investigator to be of no clinical significance are also allowed to be included).
12. For patients with reproductive potential, blood or urine pregnancy tests must be negative within one week before joining the trial. If there is a risk of pregnancy, effective contraceptive measures must be used during the entire trial treatment until 180 days after the last administration (year failure rate < 1%), for example: use of physical barrier contraceptive methods (condoms) or total abstinence. Oral, injection or implantation of hormonal contraceptives are not allowed. For women without reproductive potential, defined as:

    * Naturally entering menopause and menopause for more than 1 year.
    * Surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
    * Serum follicle stimulating hormone, luteinizing hormone and plasma estradiol levels are within the menopausal standards of the research center laboratory.
13. Patients must understand the trial process and have the ability to comply with the trial protocol within the study period, including any treatment, examination, inspection, follow-up and questionnaire required to accomplish the trial.
14. Patients must be willing to complete the quality of life questionnaires during the trial treatment and the follow-up, and agree that the results of these questionnaires will be used for clinical research.
15. Any side effects of previous chemotherapy must have returned to ≤ CTCAE level 1 or baseline level, except for sensory neuropathy or alopecia with stable symptoms ≤ CTCAE level 2.

Exclusion Criteria:

1. Personnel involved in the formulation or implementation of research plans.
2. Histological evidence of non-ovarian clear cell carcinoma.
3. Lack of tumor samples (archived and/or recently obtained).
4. Previous administration of the following therapies in the past: anti-PD-1/PD-L1/PD-L2 drugs; or anti stimulating/synergistic inhibition of T cell receptor (for example, CTLA-4, CD134, CD137) drugs.
5. Patients with contraindications of bevacizumab, including but not limited to: previous gastrointestinal perforation, receiving surgery or having incomplete-healing wound within 28 days before administration of combination therapy, severe bleeding or recent hemoptysis, and other circumstances that are inappropriate for bevacizumab according to physician's assessment.
6. Patients are known to be allergic to the active ingredients or excipients of sintilimab or bevacizumab.
7. Symptomatic or uncontrolled brain metastases that require simultaneous treatment, including but not limited to surgery, radiation and/or corticosteroids, or clinical manifestations of spinal cord compression.
8. Currently participating in interventional clinical research treatment, or received other research drugs or used research equipment treatment within 4 weeks before the first administration.
9. Diagnosis of other malignant diseases other than ovarian cancer within 5 years before the first administration (excluding radically cured skin basal cell carcinoma, skin squamous cell carcinoma, and/or radically excised carcinoma in situ).
10. An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatments a.
11. Active hemoptysis (at least 2.5ml or 1/2 teaspoon of blood was spit out at a time) within 3 months before the first administration.
12. Patients have been vaccinated with live vaccine within 1 month before the first administrationb.
13. Patients have received platelet or red blood cell transfusion within 4 weeks before the first administration.
14. Patients receive major surgery within 4 weeks before the first administration (except for surgery for the purpose of biopsy) or expect major surgery during the study period.
15. Patient have received systemic treatment with anti-tumor Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural fluid) within 2 weeks before the first administration.
16. Patients are receiving systemic glucocorticoid therapy (not including nasal spray, inhaled or other local glucocorticoids) or any other form of immunosuppressive therapy (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide and anti-TNF drugs)c.
17. Minor surgery (outpatient or inpatient surgery requiring local anesthesia, including central venous catheterization) within 48 hours before the first administration.
18. Use aspirin (>325 mg/day) or other non-steroidal anti-inflammatory drugs known to inhibit platelet function for 10 consecutive days at present or in the future (within 10 days before first administration).
19. Current or recent (within 10 days before first administration) full-dose oral or parenteral anticoagulant or thrombolytic treatment for 10 consecutive daysd.
20. Patients have a hereditary bleeding tendency or coagulation dysfunction, or a history of thrombosis. Or the image shows tumor invasion/infiltration of large blood vessels or the researchers or radiologists assess the bleeding tendency.
21. Clinically uncontrolled pleural effusion/abdominal effusion (patients who do not need to drain the effusion or stop drainage for 3 days without a significant increase in effusion can be included).
22. Severe unhealed wound ulcers or fractures.
23. Known allogeneic organ transplantation (except for corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
24. Known human immunodeficiency virus (HIV) infection history (HIV 1/2 antibody positive).
25. Untreated active hepatitis B (defined as HBsAg positive and the number of copies of HBV-DNA detected at the same time is greater than the upper limit of the normal value of the laboratory department of the research center)e.
26. Patients who are pregnant or breastfeeding, or expect to become pregnant during the study treatment period.
27. There is clinically unresolved toxicity from previous treatments (≥ Grade 2, except for alopecia, neuralgia, lymphopenia, and depigmentation of skin).
28. There are any severe or uncontrolled systemic diseases, such as:

    * The resting electrocardiogram has major abnormalities in rhythm, conduction, or morphology that are severe and difficult to control, such as complete left bundle branch block, above II degree of heart block, ventricular arrhythmia, or atrial fibrillation.
    * Unstable angina pectoris, congestive heart failure, chronic heart failure with NYHA grade ≥ 2.
    * Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack within 6 months before being selected for the trial.
    * Unsatisfactory blood pressure control (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg).
    * Active tuberculosis.
    * Active or uncontrolled infection that requires systemic treatment.
    * Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction.
    * Liver diseases such as liver cirrhosis, decompensated liver disease, acute or chronic active hepatitis.
    * Poor control of diabetes (FBG > 10 mmol/L).
    * Urine routines suggest that urine protein ≥ ++, and the 24-hour urine protein quantitative is confirmed to be > 1.0 g.

    Patients with mental disorders who cannot cooperate with treatment.
29. The medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the trial results, prevents the patients from participating in the study. The investigator believes that there are other potential risks and the patient is not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the proportion of patients with complete response(CR) and partial response(PR) assessed by the investigator in accordance with the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the time from enrollment to the first imaging disease progression or death (whichever occurs first). Assessed according to RECIST v1.1 by investigator.
Time to response (TTR) | Up to 2 years
  TTR is defined as the time from the first administration to the first CR or PR recorded. Assessed according to RECIST v1.1 by investigator.
Duration of remission (DOR) | Up to 3 years
  DOR is defined as the time interval from the first record of disease response to disease progression or death (whichever occurs first). Assessed according to RECIST v1.1 by investigator.
Disease control rate (DCR) | Up to 5 years
  DCR is defined as the proportion of the patients with complete response, partial remission, and stable disease after treatment. Assessed according to RECIST v1.1 by investigator.
Overall survival (OS) | Up to 5 years
  OS is defined as the time between enrollment and the patient's death due to any cause.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 3 years
  Safety includes the adverse event profile of sintilimab and bevacizumab according to the Common Terminology Criteria for Adverse Events version 5.0.
Quality of life assessment of patients | Quality of life will be assessed by Functional Assessment of Cancer Therapy-Ovarian (FACT-O)
  Quality of life will be assessed by Functional Assessment of Cancer Therapy-Ovarian (FACT-O) and other scales as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available (including data dictionaries). The individual participant data that underlie the results reported in this article after deidentification (text, tables, figures, and appendices) in particular will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available immediately following publication without end date.
Access Criteria: To obtain the data, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Peng Z, Li H, Gao Y, Sun L, Jiang J, Xia B, Huang Y, Zhang Y, Xia Y, Zhang Y, Shen Y, Huang B, Nie J, Chen X, Liu X, Feng C, Li Z, Zhang W, Tao K, Zhang Q, Duan S, Chen Y, Chen Y, Wang W, Zheng H, Lu Y, Liu Y, Wang L, Qi W, He Y, Tian Y; NUWA Platform Research Group; Li G, Ma D, Gao Q. Sintilimab combined with bevacizumab in relapsed or persistent ovarian clear cell carcinoma (INOVA): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2024 Oct;25(10):1288-1297. doi: 10.1016/S1470-2045(24)00437-6. Epub 2024 Sep 11. PMID 39276785
- [Derived] Li R, Liu X, Song C, Zhang W, Liu J, Jiao X, Yu Y, Zeng S, Chi J, Zhao Y, Ma G, Huo Y, Li M, Peng Z, Li G, Jiang J, Gao QL. Sintilimab combined with bevacizumab in relapsed/persistent ovarian clear cell carcinoma (INOVA): an investigator-initiated, multicentre clinical trial-a study protocol of clinical trial. BMJ Open. 2022 May 24;12(5):e058132. doi: 10.1136/bmjopen-2021-058132. PMID 35613822